CLINICAL TRIAL: NCT00380549
Title: A Prospective Case Series (Pilot Study) Comparing Ion Levels and Clinical Outcomes of the CONSERVE® A-Class Type Hip System With BFH™ Technology to the CONSERVE® Plus Total Hip Resurfacing System
Brief Title: A Comparison of an Advanced Metal Hip System to a Resurfacing Hip System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OHREB 2005884-01H
Record Dates: First submitted 2006-09-23; First posted 2006-09-26 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis, hip replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONSERVE® A-Class THA BFH (Active Comparator): CONSERVE® A-Class Total Hip with BFH technology. Patients in this arm will undergo a unilateral total hip replacement with the CONSERVE® acetabular component and the CONSERVE® A-Class BFH femoral head. Blood ion levels will be collected and analyzed.
  Interventions: Diagnostic Test: Blood ion levels
- CONSERVE® Plus Total Resurfacing Hip System (Active Comparator): CONSERVE® Plus Total Resurfacing Hip System. Patients in this arm will undergo a unilateral total hip replacement with the CONSERVE® Plus Total Resurfacing Hip System. Blood ion levels will be collected and analyzed.
  Interventions: Diagnostic Test: Blood ion levels

INTERVENTIONS:
Diagnostic Test: Blood ion levels — Blood ion levels or the levels of cobalt and chromium ions in the blood and urine will be analyzed.

SUMMARY:
The primary purpose of the current study is to investigate if the CONSERVE® A-Class Total Hip with BFH technology will lead to lower blood ion levels in patients, as compared to patients in a recent study who received the CONSERVE® Plus Total Resurfacing Hip System, another metal-on-metal device. We are also comparing functional and radiographic (x-rays) outcomes between patients who receive the CONSERVE® A-Class Total Hip compared to those who have received the CONSERVE® Plus Total Resurfacing Hip System.

DETAILED DESCRIPTION:
A standard hip replacement involves replacing your hip joint with several parts: the cup which forms the socket in the pelvis; a head that forms a new ball for the top of the thigh bone; and a stem which is placed into the thigh bone. Typically, the socket is made out of metal and plastic, and the ball and stem are made out of metal.

Recently, new metal-on-metal hip replacement systems have been developed where both the socket and the shell are made out of metal. This can cause metal ions to be released into the body. The CONSERVE® A-Class Total Hip with BFH technology is a new metal-on-metal total hip system which utilizes a large diameter femoral head (36-54 mm) more similar to the size of the original head (i.e., your original bone). Further, this system utilizes an advanced metal design which wears at a slower rate than typical metal-on-metal implants. Therefore, the primary purpose of the current study is to investigate if the CONSERVE® A-Class Total Hip with BFH technology will lead to lower blood ion levels in patients, as compared to patients in a recent study who received the CONSERVE® Plus Total Resurfacing Hip System, another metal-on-metal device. We are also comparing functional and radiographic (x-rays) outcomes between patients who receive the CONSERVE® A-Class Total Hip compared to those who have received the CONSERVE® Plus Total Resurfacing Hip System.

ELIGIBILITY:
Inclusion Criteria:

* (1) Individuals undergoing unilateral total hip replacement with the CONSERVE® acetabular component and the CONSERVE® A-Class BFHä femoral head in combination with an uncemented femoral stem produced from the Ti-6A1-4V alloy (ASTM F-136) with or without titanium plasma coating.

  (2) Patients who are undergoing primary hip surgery for Noninflammatory Degenerative Joint Disease (NIDJD). Composite diagnoses of NIDJD include osteo/degenerative arthritis, traumatic arthritis, congenital hip dysplasia, and avascular necrosis.

  (3) Patients 18 years of age or older (skeletally mature). (4) Patients for whom there is a reasonable expectation that they will be available for each examination scheduled over a two year post-operative follow-up period and for annual exams until the last patient entered into the study has achieved two years of follow-up.

  (5) Patients who agree to participate and sign the Informed Consent Form. (6) Patients who do not meet any of the exclusion criteria.

Exclusion Criteria:

* (1) Patients with previous fusions, acute femoral neck fractures, above knee amputations, or significant arthritic changes to the knees.

  (2) Patients with evidence of active infection. (3) Patients with neurologic or musculoskeletal disease that may adversely affect gait or weight-bearing.

  (4) Patients who have previously undergone an ipsilateral hemi resurfacing, total resurfacing, total bipolar, unipolar or total hip replacement device.

  (5) Patients with neuropathic joints. (6) Patients with severe documented psychiatric disease. (7) Patients requiring structural bone grafts. (8) Patients with a documented allergy to cobalt chromium molybdenum. (9) Patients with an ipsilateral girdlestone. (10) Patients with sickle cell disease. (11) Patients with renal failure as defined by serum creatinine level greater than 180 Fmol/L.

  (12) Patients who otherwise meet the study criteria, but refuse to consent in writing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
blood ion levels | 2 years post-operative
  Assessment of Chromium and Cobalt ion levels in the blood

SECONDARY OUTCOMES:
functional outcomes radiographic outcomes complication rates | 2 years post-operatively
  Assessment of clinical efficiency of the implant by validated questionannires and radiographic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kim, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Beaule PE, Kim PR, Hamdi A, Fazekas A. A prospective metal ion study of large-head metal-on-metal bearing: a matched-pair analysis of hip resurfacing versus total hip replacement. Orthop Clin North Am. 2011 Apr;42(2):251-7, ix. doi: 10.1016/j.ocl.2011.01.005. PMID 21435499